CLINICAL TRIAL: NCT05432791
Title: A Randomized Phase 2/3 Study of Olaparib Plus Temozolomide Versus Investigator's Choice for the Treatment of Patients With Advanced Uterine Leiomyosarcoma After Progression on Prior Chemotherapy
Brief Title: Testing Olaparib and Temozolomide Versus the Usual Treatment for Uterine Leiomyosarcoma After Chemotherapy Has Stopped Working
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-05065; NCI-2022-05065 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A092104 (Other: Alliance for Clinical Trials in Oncology); A092104 (Other: CTEP); U10CA180821 (NIH); NCT05633381 (obsolete NCT alias)
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Uterine Corpus Leiomyosarcoma; Metastatic Uterine Corpus Leiomyosarcoma; Stage III Uterine Corpus Leiomyosarcoma AJCC v8; Stage IV Uterine Corpus Leiomyosarcoma AJCC v8; Unresectable Uterine Corpus Leiomyosarcoma
MeSH Terms: interventions — Specimen Handling; Magnetic Resonance Spectroscopy; olaparib; pazopanib; Temozolomide; Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (olaparib, temozolomide) (Experimental): Patients receive temozolomide PO QD on days 1-7 of each cycle and olaparib PO BID on days 1-7 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan or MRI and/or bone scans throughout the trial. Patients also undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Olaparib; Drug: Temozolomide; Procedure: Transthoracic Echocardiography Test
- Arm 2 (trabectedin, pazopanib) (Active Comparator): Patients receive trabectedin IV continuously over 24 hours on day 1 of each cycle or pazopanib PO QD on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan or MRI and/or bone scans throughout the trial. Patients also undergo TTE or MUGA on study and as clinically indicated, as well as collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Pazopanib; Drug: Trabectedin; Procedure: Transthoracic Echocardiography Test

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
  Arms: Arm 1 (olaparib, temozolomide)
Drug: Pazopanib — Given PO
  Other Names: GW786034
  Arms: Arm 2 (trabectedin, pazopanib)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
  Arms: Arm 1 (olaparib, temozolomide)
Drug: Trabectedin — Given IV
  Other Names: Ecteinascidin; Ecteinascidin 743; ET 743; ET-743; ET743; Yondelis
  Arms: Arm 2 (trabectedin, pazopanib)
Procedure: Transthoracic Echocardiography Test — Undergo TTE
  Other Names: TRANSTHORACIC ECHOCARDIOGRAPHY; TTE

SUMMARY:
This phase II/III trial compares the effect of the combination treatment with olaparib and temozolomide to trabectedin or pazopanib (two of the most common chemotherapy drugs used as usual approach) in patients with uterine leiomyosarcoma that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) after initial chemotherapy has stopped working. The usual approach is defined as care most people get for advanced uterine leiomyosarcoma. Olaparib is a PARP inhibitor. PARP is a protein that helps repair damaged deoxyribonucleic acid (DNA). Blocking PARP may prevent tumor cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. Temozolomide is in a class of medications called alkylating agents. It works by slowing or stopping the growth of tumor cells in the body. The combination of olaparib and temozolomide may work better than the usual treatment in shrinking or stabilizing advanced uterine leiomyosarcoma after initial chemotherapy has stopped working.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression free survival (PFS) of olaparib plus temozolomide (Arm 1) as compared to investigator's choice (trabectedin or pazopanib hydrochloride [pazopanib]) (Arm 2) for the treatment of patients with advanced uterine leiomyosarcoma (uLMS) who have received two or more prior lines of therapy as determined by investigator (local site) assessment. (Phase 2) II. To compare the overall survival (OS) of olaparib plus temozolomide (Arm 1) as compared to investigator's choice (trabectedin or pazopanib) (Arm 2) for the treatment of patients with advanced uLMS who have received two or more prior lines of therapy. (Phase 3)

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of each treatment by determining adverse events using Common Terminology Criteria for Adverse Events (CTCAE) version 5 and patient-reported toxicity using Patient-Reported Outcome (PRO)-CTCAE version 1 in and across each treatment arm. (Phase 2/3) II. To evaluate the objective response rate (ORR), duration of response (DOR) and disease control rate (DCR) in and across each treatment arm as determined by investigator assessment. (Phase 2/3)

EXPLORATORY OBJECTIVE:

I. To collect results of tumor genomic testing previously conducted as part of clinical care (when available) and (a) to determine the proportion of patients with a genomic alteration in a homologous recombination (HR) pathway gene and (b) to evaluate for any relationship between the presence of such an alteration and clinical benefit from olaparib and temozolomide. (Phase 2/3)

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive temozolomide orally (PO) once daily (QD) on days 1-7 of each cycle and olaparib PO twice daily (BID) on days 1-7 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan or magnetic resonance imaging (MRI) and/or bone scans throughout the trial. Patients also undergo collection of blood samples throughout the trial.

ARM 2: Patients receive trabectedin intravenously (IV) continuously over 24 hours on day 1 of each cycle or pazopanib PO QD on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan or MRI and/or bone scans throughout the trial. Patients also undergo transthoracic echocardiography (TTE) or multi-gated acquisition scan (MUGA) on study and as clinically indicated, as well as collection of blood samples throughout the trial.

After completion of study treatment, patients without disease progression are followed every 6 weeks until disease progression. After disease progression, patients are followed every 3 months for the first 2 years, then every 6 months thereafter until 5 years post-randomization or death, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed leiomyosarcoma of uterine origin, as established by the site institutional practice for pathology confirmation for research studies when enrolling the patient on study. Central pathology review will not occur.
* Metastatic or locally advanced and surgically unresectable disease, in the opinion of the treating investigator.
* Patients must have at least one lesion that is measurable per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria to be eligible for the study.
* Not pregnant and not nursing, because this study involves agents that have known genotoxic, mutagenic and teratogenic effects. Therefore, for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required
* Age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status =< 2.
* Patients must have had prior progression on, or intolerance to, at least two prior lines of systemic therapy for advanced uLMS, one of which was an anthracycline (anthracycline monotherapy or combination). Adjuvant chemotherapy will qualify as a prior line of treatment. Endocrine treatment will not qualify as a prior line of treatment.
* Patients may not have received prior treatment with any PARP inhibitor, temozolomide or dacarbazine (IV analogue of temozolomide).
* Patients may not have had prior treatment with BOTH of the agents included on the investigator's choice arm: trabectedin AND pazopanib. If the patient has had prior treatment with one of these agents, they are eligible; however, they must be assigned to the other agent for investigator's choice. That is, patients who have received prior pazopanib must be assigned to trabectedin, and patients who have received prior trabectedin must be assigned to pazopanib.
* Patients must have recovered to baseline or =< grade 1 per CTCAE version 5.0 from toxicity related to any prior treatment, unless adverse events are clinically nonsignificant and/or stable on supportive therapy, with the exception of fatigue (which must be =< grade 2), alopecia and/or endocrinopathies related to prior immunotherapy which are controlled with hormone replacement.
* Patients must have completed all prior anti-cancer treatment, including radiation, >= 28 days prior to registration.
* Patients may have undergone major surgery (related or unrelated to their cancer diagnosis) >= 28 days of registration. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* Absolute neutrophil count (ANC) >= 1500/mm^3 (within =< 28 days prior to registration).
* Platelet count >= 100,000/mm^3 (within =< 28 days prior to registration).
* Creatinine =< 1.5 * upper limit of normal (ULN) (within =< 28 days prior to registration).

  * If creatinine > 1.5 * ULN, then creatinine clearance (CrCl) must be > 50 mL/min, per Cockcroft-Gault method.
* Hemoglobin >= 9 g/dL (within =< 28 days prior to registration).

  * No transfusions =< 14 days before cycle 1 day 1 (C1D1).
* Total bilirubin =< 1.5 x ULN (within =< 28 days prior to registration).

  * If documented Gilbert's: =< 2.0 x ULN.
* Aspartate aminotransferase/alanine aminotransferase (AST/ALT) =< 3 x ULN (within =< 28 days prior to registration).
* Patients may not have uncontrolled hypertension defined as a blood pressure (BP) > 150/90 on two consecutive assessments during the screening period. If a patient is found to have a BP > 150/90 on two consecutive assessments during the screening period, the patient may be started on an anti-hypertensive regimen, and will be considered eligible if two subsequent measurements are performed and the BP is =< 150/90. If BP is in range on the first measurement, no further measurements are needed.
* Patients must demonstrate a QTcF (Fredericia formula) =< 470 msec on an electrocardiography (EKG) performed during screening. This criterion applies only to patients who will receive pazopanib if randomized to Arm 2. Repeat EKG testing during the screening period is allowed.
* Patients may not have an uncontrolled ventricular arrhythmia or recent (within 3 months) myocardial infarction.
* In addition to the above, patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible, patients should be class 2B or better.
* Patients may not have a history of active or unresolved: perforation, abscess or fistula within 28 days prior to registration (either clinically or radiographically).
* Patients must not have myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or a history of bone marrow biopsy findings at any time consistent with MDS and/or AML.
* For patients with evidence of chronic hepatitis B (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with central nervous system (CNS)/leptomeningeal disease must have undergone definitive treatment, have no evidence of CNS progression on follow-up imaging performed at least 4 weeks after the CNS-directed therapy is completed, and be off all steroids, in order to be eligible.
* Patients must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any other condition that would limit compliance with study requirements.
* Patients must be able to swallow oral medications.
* Patients may not require concomitant use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks.
* Patients may not require concomitant use of known strong (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* In order to complete the mandatory patient-completed measure, participants must be able to speak and/or read English and Spanish. Non-English or non-Spanish readers may still participate in the study but are not required to complete the PRO-CTCAE side effect surveys.
* For all patients, prior to randomization and as part of eligibility, the investigator must select the agent which the patient would receive if assigned to the investigator's choice arm, prior to randomization. The patient must meet all eligibility criteria for that agent during screening and prior to randomization.
* Patients without central venous access must be willing to undergo placement of central venous access (i.e. port or peripherally inserted central catheter [PICC] line, per institutional practice) if assigned to the investigator's choice arm and if the investigator intends to treat the patient with trabectedin. The site must be able to place central venous access within 10 days of registration/randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) (Phase II) | Time between the date of randomization and the earliest of disease progression or death, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method, where the stratified log-rank test will be used to compare the distributions across the treatment arms. PFS rates at 1 year, 2 years, and 5 years will also be reported, along with 95% confidence intervals. Univariable and multivariable Cox models stratified by the stratification factors used in the randomization will be assessed as well.
Overall survival (OS) (Phase III) | Time between the date of randomization and the date of death from any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method, where the stratified log-rank test will be used to compare the distributions across the treatment arms. OS rates at 1 year, 2 years, and 5 years will also be reported, along with 95% confidence intervals. Univariable and multivariable Cox models stratified by the stratification factors used in the randomization will be assessed as well.

SECONDARY OUTCOMES:
Overall response rate | Up to 5 years
  Will be estimated by dividing the number of evaluable patients that achieve a confirmed response (partial response [PR] or better) by the total number of evaluable patients. This estimate will be calculated by arm and will also include a 95% confidence interval using the properties of the binomial distribution, and compared between the arms using a chi-square test.
Duration of response (DOR) | Time from first evidence of response until disease progression (or death), assessed up to 5 years
  This analysis is restricted to those patients that achieved a confirmed response (PR or better). Patients that go off of study treatment prior to progression will have their DOR time censored at that time.
Disease control rate | Up to 6 weeks
  Will be estimated using the number of patients that achieve complete response, partial response, or stable disease at the 6 week assessment divided by all evaluable patients. This estimate will be calculated by arm and will also include a 95% confidence interval using the properties of the binomial distribution, and compared between the arms using a chi-square test.
Incidence of adverse events | Up to 4 weeks after the end of study treatment
  Adverse events will be recorded using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for each patient. Frequency tables and summary statistics will be used and with the appropriate methods of evaluating categorical and continuous data. In addition, patient reported safety and tolerability will be assessed using Patient-Reported Outcomes (PRO)-CTCAE for a prespecified group of expected toxicities. PRO-CTCAE assessments will occur prior to registration and on day 1 of every cycle during treatment. Collection of PRO-CTCAE will be discontinued after cycle 11.

OTHER OUTCOMES:
Proportion of patients with a genomic alteration in a homologous recombination (HR) pathway gene | Within 60 days of registration
  Will collect results of next generation sequencing that is known to the treating investigator and was previously performed as part of the patient's clinical care, for all patients registered to the study. Will evaluate for genomic alterations in HR pathway genes. A genomic alteration is defined as a homozygous deletion or deleterious (loss-of-function) mutation in any of the pre-defined HR pathway genes.
Relationship between the presence of an alteration in HR pathway genes and clinical benefit from olaparib and temozolomide | Assessed up to 5 years
  Will evaluate whether patients with an HR pathway alteration experience increased clinical benefit from olaparib and temozolomide as compared patients who lack such an alteration, as determined by objective response rate, progression-free survival and overall survival. Response rates will be compared using the Fisher's exact test, and time to event endpoints summarized using the Kaplan-Meier curves and the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ingham, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (145):
- United States (144):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - Our Lady of the Lake Medical Oncology, Baton Rouge, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - ECU Health Medical Center, Greenville, North Carolina
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Centro Comprensivo de Cancer de UPR, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT05432791/ICF_000.pdf